CLINICAL TRIAL: NCT04109781
Title: Short Clinical Outcome of Microscope Assisted Discectomy: Results of 90 Cases in Iraq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan2
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: To Evaluate the Effectiveness if Microscope in Discectomy
Keywords: short-term clinical outcome; microscopic assisted discectomy; lumbar disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Lumbar disc herniation (Other): Patients with lumbar disc herniation with no response to conservative treatment and were treated with Microdiscectomy
  Interventions: Procedure: Microscope assisted discectomy

INTERVENTIONS:
Procedure: Microscope assisted discectomy — Microdiscectomy

SUMMARY:
A total of (90) patients involved in this study a randomized sampling use. The adult patient between (17) and (50) years of age complaining of lower back pain; and or radiculopathy and neurological symptoms, whom failed to respond to a (6-8) weeks period of conservative therapy (life style modification, NSAIDs, and physiotherapy). They are operated by Microscopic assisted discectomy and were followed by ODI and VAS for back pain and leg pain for 4 months after surgery

DETAILED DESCRIPTION:
A total of (90) patients involved in this study a randomized sampling use. The adult patient between (17) and (50) years of age complaining of lower back pain; and or radiculopathy and neurological symptoms, whom failed to respond to a (6-8) weeks period of conservative therapy (life style modification, NSAIDs, and physiotherapy). The diagnosis carried out using history, physical examination, MRI done for the patient to confirm the diagnosis and the level of disc herniation and know the direction and extend of disc herniation.Population excluded from study were the age group above or less the ones whom involved in the study, any other type of disc herniation apart from L3-L4, L4-L5, L5-S1, multilevel pathology, patients with spondylolisthesis, spondylolysis, patients with scoliosis and kyphosis, patients with cauda equina syndrome, patients with previous back surgery, and with no local infection.All the patients discharged on the same day of operation or a day after, mobilized soon as they were ready. Patient were reviewed in intervals of (2) weeks (2) months and (4) months after surgery using VAS for low back pain and leg pain and Oswestry disability index.

ELIGIBILITY:
Inclusion Criteria:

* lower back pain; and or radiculopathy and neurological symptoms, whom failed to respond to a (6-8) weeks period of conservative therapy (life style modification, NSAIDs, and physiotherapy).

Exclusion Criteria:

* Population excluded from study were the age group above or less the ones whom involved in the study, any other type of disc herniation apart from L3-L4, L4-L5, L5-S1, multilevel pathology, patients with spondylolisthesis, spondylolysis, patients with scoliosis and kyphosis, patients with cauda equina syndrome, patients with previous back surgery, and with no local infection.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue score for back and leg pain | Visual analogue score was assessed in all patients preoperatively and then assessed postoperatively at 2 weeks , 2 months and 4 months which showed that there is changes after operation which indicates improvement by Microdiscectomy
  Visual analogue score for back pan and leg pain is measurement of patient feeling of pain which can be from 0 (no pain) to 10 ( severe pain )
Oswestry disability index | Oswestry disability index was assessed preoperatively and postoperatively at 2 weeks , 2 months and 4 months and showed there is improvement in this index after surgery which indicates improvement with microdiscecetomy
  Oswestry disability index is low back pain questionnaire as followingFor each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) 50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated: 16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement)